CLINICAL TRIAL: NCT05871021
Title: A Phase IIa, Open-label, Multicenter Study of Radiochemotherapy With Isotoxic Dose Escalation and Protective VEGF Inhibition Using Bevacizumab in the Treatment of Patients With First Diagnosis of IDH Wild-type, MGMT Unmethylated Glioblastoma
Brief Title: Protective VEGF Inhibition for Isotoxic Dose Escalation in Glioblastoma
Acronym: PRIDE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-000565-32
Record Dates: First submitted 2023-04-30; First posted 2023-05-23 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-09

CONDITIONS: Glioblastoma
Keywords: Dose escalation; bevacizumab; VEGF inhibition; FET PET; VMAT
MeSH Terms: conditions — Glioblastoma | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 75 Gy with two cycles of bevacizumab (Experimental)
  Interventions: Radiation: Dose escalation of radiation dose beyond the therapeutic standard

INTERVENTIONS:
Radiation: Dose escalation of radiation dose beyond the therapeutic standard — Dose escalation to 75 Gy with concomitant radioprotectant bevacizumab
  Other Names: bevacizumab

SUMMARY:
Glioblastoma is the most aggressive brain tumor and often recurs locally despite intensive treatment. Standard chemoradiotherapy with 60 Gy may not be sufficient to control the tumor, and dose escalation seems to be warranted, but causes more toxicity. To address this, the multicentric PRIDE trial employs two cycles of bevacizumab to achieve dose escalation isotoxically. The goal is improved survival without significantly increasing side effects. The study uses a simultaneous integrated boost with a total dose of 75 Gy in 2.5 Gy per fraction.

ELIGIBILITY:
Inclusion Criteria:

* IDH wild-type, MGMT unmethylated glioblastoma patients
* Informed consent
* Age ≥18 and ≤70 years, smoking or non-smoking, of any ethnic origin
* ECOG 0-2
* Neutrophil counts >1500/µl, Platelet counts >100.000/µl, Hemoglobin > 8 g/dl, Serum creatinine <1.5-fold upper limit of normal (ULN), Bilirubin, AST or ALT <2.5-fold ULN unless attributed to anticonvulsants, Alkaline phosphatase <2.5-fold ULN
* Adequate contraception
* Serum creatinine ≤ 1.5 x ULN AND patients with urine dipstick for proteinuria < 2+. Patients with ≥ 2+ proteinuria on dipstick urinalysis at baseline should show urine protein to creatinine ratio ≤ 1

Exclusion Criteria:

* Evidence of significant hemorrhage on postoperative MRI of the brain. Patients with asymptomatic, minor hemosiderin deposition, resolving postsurgical hemorrhagic changes, or punctate intratumoral hemorrhage (e.g., related to biopsy or surgery) are not excluded
* Subjects on any drug suspected to interfere with bevacizumab at the time of study inclusion
* Immuno-compromised patients, including known seropositivity for human immunodeficiency virus (HIV)
* Known hypersensitivity to any component of the investigational drugs or excipients (allergy to or other intolerability of bevacizumab or excipients)
* Any other significant medical illness or medically significant laboratory finding that would, in the investigator's judgement, make the patient inappropriate for this study, or would increase the risk associated with the patients' participation in the study
* Incapability to undergo MRI
* Prior treatment with bevacizumab for any indication
* Contraindication and/or hypersensitivity to bevacizumab or its excipients. For details check the Summary of Product Characteristics Aybintio®
* Significant cardiovascular disease defined as congestive heart failure (NYHA Class II, III, IV), unstable angina pectoris, or myocardial infarction within 6 months prior to enrolment
* Inadequately controlled hypertension (defined as a blood pressure of > 150 mmHg systolic and/or >100 mmHg diastolic on medication), or any prior history of hypertensive crisis or hypertensive encephalopathy
* History of clinically significant cerebrovascular events within 6 months prior to enrolment. This includes ischemic stroke or transient ischemic attack. Small, clinically silent perioperative ischemic changes are not exclusionary.
* Significant vascular disease (e.g. aortic aneurysm, aortic dissection or recent peripheral arterial thrombosis) within 6 months prior to enrolment
* Evidence or history of recurrent thromboembolism (> 1 episode of deep venous thrombosis / peripheral embolism) during the past 2 years
* Evidence of bleeding diathesis or coagulopathy (in the absence of therapeutic anticoagulation)
* Chronic daily intake of aspirin > 325 mg/day or clopidogrel > 75 mg /day
* History of intracranial abscess within 6 months prior to inclusion
* History of abdominal or tracheo-oesophageal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to study enrolment
* History of ≥ grade 2 hemoptysis according to NCI-CTC criteria within 1 month prior to inclusion
* Serious non-healing wound, ulcer or bone fracture

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2024-04-10 (Actual); Primary Completion 2028-04-10 (Estimated); Study Completion 2028-07-10 (Estimated)

PRIMARY OUTCOMES:
OS | Date of study inclusion (informed consent) to death or end of F/U
  Overall Survival

SECONDARY OUTCOMES:
Safety and tolerability | Date of study inclusion (informed consent) to death or end of F/U
  Safety and tolerability of dose escalation with bevacizumab according to CTCAE v5.0
PFS-6 | 6 months after the date of study inclusion (informed consent)
  6 months rate of progression-free survival
PFS | Date of study inclusion (informed consent) to death or progression
  Progression-free survival
QoL | Date of study inclusion (informed consent) to death or end of F/U
  Quality of life as determined by EORTC QLQ-C30/QLQ-BN 20
Cognitive function | Date of study inclusion (informed consent) to death or end of F/U
  Cognitive function determined by standard test batteries
Exploratory objective | Date of study inclusion (informed consent) to death or end of F/U
  Validation of prognostic 4-miRNA signature-based risk score

CONTACTS AND LOCATIONS:
Overall Officials: Maximilian Niyazi, Prof. Dr., Principal Investigator — University Hospital Tuebingen, Department of Radiation Oncology
Locations (1):
- Department of Radiation Oncology, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maier SH, Schonecker S, Anagnostatou V, Garny S, Nitschmann A, Fleischmann DF, Buttner M, Kaul D, Imhoff D, Fokas E, Seidel C, Hau P, Kolbl O, Popp I, Grosu AL, Haussmann J, Budach W, Celik E, Kahl KH, Hoffmann E, Tabatabai G, Paulsen F, Holzgreve A, Albert NL, Mansmann U, Corradini S, Belka C, Niyazi M, Bodensohn R. Dummy run for planning of isotoxic dose-escalated radiation therapy for glioblastoma used in the PRIDE trial (NOA-28; ARO-2024-01; AG-NRO-06). Clin Transl Radiat Oncol. 2024 May 4;47:100790. doi: 10.1016/j.ctro.2024.100790. eCollection 2024 Jul. PMID 38765202
- See also: Dosimetric feasibility analysis and presentation of an isotoxic dose-escalated radiation therapy concept for glioblastoma used in the PRIDE trial — https://pubmed.ncbi.nlm.nih.gov/38116137/
- See also: Dummy run for planning of isotoxic dose-escalated radiation therapy for glioblastoma used in the PRIDE trial (NOA-28; ARO-2024-01; AG-NRO-06) — https://pubmed.ncbi.nlm.nih.gov/38765202/
- See also: FET PET-based target volume delineation for the radiotherapy of glioblastoma: A pictorial guide to help overcome methodological pitfalls — https://pubmed.ncbi.nlm.nih.gov/38880414/